CLINICAL TRIAL: NCT05509179
Title: Evaluation of the Implementation of Neonatal Phototherapy With BiliCocoon® in Maternity Wards
Acronym: BiliCocoon
Status: Completed | Type: Observational
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Other Study IDs: BiliCocoon
Record Dates: First submitted 2022-08-18; First posted 2022-08-22 (Actual); Last update posted 2023-04-27 (Actual); Status verified 2023-04

CONDITIONS: Neonatal Phototherapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Free bilirubin jaundice is a common condition in the neonatal period: 80% of newborns have some degree of hyperbilirubinemia within days of birth, but only 5-10% require treatment to prevent complications or to treat the cause of jaundice. The major complication is neurological toxicity, the most severe form of which is kernicterus, a severe and irreversible hyperbilirubinemic encephalopathy involving the basal ganglia. The main treatment for jaundice is phototherapy, which may or may not be combined with exchange transfusion in the most severe forms of jaundice caused by uncontrolled severe hemolysis. Phototherapy acts by interaction of light with bilirubin located in the skin, transforming it into photo-derivatives directly eliminated in the stool and urine. The hepatic stage of bilirubin transformation, limiting its elimination in newborns, is thus short-circuited. The interaction between bilirubin and light on the skin is maximal in the 460-490 nm spectrum. Phototherapy technology has evolved considerably since the discovery of its effectiveness by Dr. Cremer in 1958, with a constant progression in its effectiveness and indications. The light sources used in phototherapy devices are varied and today all use Light Emitting Diode (LED) technology. The models used today in phototherapy directly emit a blue wavelength, whose spectrum between 420 and 490 nm is the most effective. The effectiveness of the treatment also depends on the exposed skin surface, the homogeneity of the light intensity and the distance between the skin and the light source.

Other phototherapy equipment is also available, including the BiliCocoon® (Bilicocoon Bag, Eurocare®). This is a so-called "proximity" equipment. Thanks to the routing of the luminous flux by an optical fiber, the terminal light panel is put directly in contact with the baby's skin. This device allows an intensive and homogeneous radiation (35 µW/cm²/nm), and a wide coverage of the body surface (1200 cm²). The Bilicocoon® is a safe and controlled therapy that is performed in the mother's room, thus avoiding any separation, allows, during the treatment, to continue breastfeeding, is easy to install, does not require goggles and therefore no scope or hospitalization and thus reduces the workload of the nursing staff. A continuous treatment of 12 hours is required, interrupted only for the baby's change. Several sessions are sometimes necessary, and in case of failure, the child can be put under intensive phototherapy. The BiliCocoon® was implemented in our maternity hospital in August 2020 to avoid mother-child separations and to limit the number of hospitalizations in neonatology.

The objective of our study is to evaluate the impact on the number of hospitalizations in neonatology since its implementation, the failure rate (unchanged or increased bilirubinemia at the end of the Bilicocoon® session requiring a relai by intensive phototherapy) and the average length of stay of neonates treated for jaundice in the NDBS maternity unit of the GHPSJ. The secondary objectives are to evaluate the failure rate of Bilicocoon® : need for intensive phototherapy after a Bilicocoon® session (Bilicocoon® failure is defined by an unchanged or increased bilirubinemia at the end of the 12-hour session) and to evaluate the length of stay of children who had Bilicocoon® alone or intensive phototherapy alone for the same causes.

ELIGIBILITY:
Inclusion Criteria:

* Newborn between 36 and 42 SA born between 01/08/2020 and 31/01/2022 at NDBS maternity
* AND in postpartum care with their mother, treated with phototherapy
* French speaking parents

Exclusion Criteria:

* Parents objecting to participation in the study
* Parents deprived of liberty
* Parents under guardianship or curatorship
* Children initially hospitalized in neonatology from the time of birth, regardless of the cause.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Newborn between 36 and 42 SA born between 01/08/2020 and 31/01/2022 at NDBS maternity and in postpartum care with their mother, treated with phototherapy
Sampling Method: Non-Probability Sample
Enrollment: 322 (Actual)
Dates: Start 2022-05-17 (Actual); Primary Completion 2022-06-17 (Actual); Study Completion 2023-04-26 (Actual)

PRIMARY OUTCOMES:
Number of hospitalizations in neonatology for free bilirubin jaundice since the introduction of Bilicocoon | Month 1
  This outcome corresponds to the number of children hospitalized in neonatology for intensive phototherapy/number of children treated for jaundice.

SECONDARY OUTCOMES:
Failure rate of Bilicocoon | Month 1
  This outcome corresponds to the number of children put under intensive phototherapy after BiliCocoon.
Length of stay of children who received Bilicocoon alone or intensive phototherapy alone | Month 1
  This outcome corresponds to the average length of stay for children treated with intensive phototherapy alone or BiliCocoon alone for the same etiology.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth WALTER, MD, Principal Investigator — Fondation Hôpital Saint-Joseph
Locations (1):
- Groupe Hospitalier Paris Saint-Joseph, Paris, France

REFERENCES:
- [Background] Luciano R, Mancini G, Cota F, Romano A, Purcaro V, Lerro F, Corsello M, Vento G. New high intensity fibreoptic phototherapy devices in healthy newborns: a single pad wrapped around the neonate body in comparison with a double pad device. Ital J Pediatr. 2019 Jun 6;45(1):68. doi: 10.1186/s13052-019-0663-5. PMID 31171028
- [Background] Bhutani VK; Committee on Fetus and Newborn; American Academy of Pediatrics. Phototherapy to prevent severe neonatal hyperbilirubinemia in the newborn infant 35 or more weeks of gestation. Pediatrics. 2011 Oct;128(4):e1046-52. doi: 10.1542/peds.2011-1494. Epub 2011 Sep 26. PMID 21949150
- [Background] Mills JF, Tudehope D. Fibreoptic phototherapy for neonatal jaundice. Cochrane Database Syst Rev. 2001;2001(1):CD002060. doi: 10.1002/14651858.CD002060. PMID 11279748
- See also: Neonatal jaundice causes and management — https://www.ijcmph.com/index.php/ijcmph/article/view/3952